CLINICAL TRIAL: NCT00199069
Title: Multicenter Trial for Treatment of Acute Lymphoblastic Leukemia in Adults (05/93)
Brief Title: German Multicenter Trial for Treatment of Newly Diagnosed Acute Lymphoblastic Leukemia in Adults (05/93)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Nicola Goekbuget, Study Coordinator, Goethe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMALL09
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Adult Acute Lymphocytic Leukemia
Keywords: ALL; Treatment; De Novo; Adult
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Vincristine; Daunorubicin; Doxorubicin; Cyclophosphamide; Ifosfamide; Cytarabine; Mitoxantrone; Methotrexate; Mercaptopurine; Thioguanine; Teniposide; Dexamethasone; Prednisolone; Stem Cell Transplantation

INTERVENTIONS:
Drug: Asparaginase
Drug: Vincristine
Drug: Daunorubicin, Adriamycin
Drug: Cyclophosphamide
Drug: Ifosfamide
Drug: Cytarabine
Drug: Mitoxantrone
Drug: Methotrexate
Drug: 6-Mercaptopurine
Drug: 6-Thioguanine
Drug: VM26
Drug: Dexamethasone / Prednisolone
Procedure: CNS Irradiation
Procedure: Mediastinal Irradiation
Procedure: Stem Cell Transplantation

SUMMARY:
The study evaluates the efficacy and tolerability of a risk- and subtype-adapted chemotherapy over one year, followed by randomized either intensified or conventional maintenance therapy. It includes a distinct protocol for the subgroup 'mature B-ALL',

ELIGIBILITY:
Inclusion Criteria:

* Acute Lymphocytic Leukemia
* Age 15 - 65 years

Exclusion Criteria:

* Serious secondary diseases which may compromise intensified chemotherapeutical treatment
* Serious psychiatric diseases, which may compromise compliance with therapy
* HIV-1 or HIV-2 Infection
* Pretreatment > 2 weeks or chemotherapy other than Vincristine and Steroids
* Patients without central diagnosis who cannot be allocated to a risk group

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 720
Dates: Start 1993-04 (Actual); Primary Completion 1999-01 (Actual); Study Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
remission rate, disease free survival, overall survival

SECONDARY OUTCOMES:
death in induction, toxicity, time and dose compliance

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hoelzer, MD, PhD, Study Chair — University of Frankfurt, Medical Department II
Locations (1):
- University Hospital, Medical Dept. II, Frankfurt, Germany

REFERENCES:
- See also: German Leukemia Trial Registry — http://www.studienregister-online.de